CLINICAL TRIAL: NCT04589858
Title: Efficacy of Specified Manual Therapies in Combination With a Supervised Exercise Protocol on Managing Pain Intensity and Functional Disability in Patients With Knee Osteoarthritis
Brief Title: Effect of Manual Therapies With Supervised Exercise Protocol on Pain and Functional Disability in Patients With Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2019-20
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Knee Osteoarthritis
Keywords: Specified manual therapy; Strengthening exercise; Stretching exercise; Knee OA; NPRS; WOMAC
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Two-arm parallel groups randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Received a supervised exercise protocol including both strengthening and stretching exercises for specific muscle groups.
  Interventions: Other: Supervised exercise protocol
- Group B (Experimental): Received manual therapies including both myofascial mobilization and manipulation technique in addition to a supervised exercise protocol.
  Interventions: Other: Supervised exercise protocol; Other: Specified Manual Therapies

INTERVENTIONS:
Other: Supervised exercise protocol — Strengthening exercises:It included a sets/group of exercises such as a static quad set in knee extension, standing terminal knee extension, seated leg-press, partial squats weight-lessened with arm support as needed, and step-ups Stretching Exercises:A slow, sustained stretching was performed in different positions for different group of muscles with holding time 30-seconds, a gap of 1-minute between two repetitions, and repeated 3-times per session on alternate day for 2-weeks. The stretching performed for the calf muscle, hamstring muscle, and quadriceps femoris muscle in standing, supine, and prone positions respectively.
Other: Specified Manual Therapies — Myofascial Mobilization: Patellar glide performed in all available ROM and direction such as superior-inferior and lateral-medial translation/glides of patella over patellar fossa.
  Myofascial manipulation technique: Manipulation of knee joint. An impulse type thrust was delivered, directed in the caudal direction to mobilize the joint in a near-full extension position.
  Arms: Group B

SUMMARY:
Osteoarthritis (OA) is referred to a group of conditions that involve mostly the larger weight-bearing joints such as the hip, knee, and ankle. It is the result of an intricate, multifaceted, progressive softening and break-down of articular cartilage along with capsular fibrosis and re-growth of new cartilages and bones called osteophytes at the margin of the articular surfaces to increase the surface area of them.

The current study aimed to find out the efficacy of specified manual therapies in combination with a supervised exercise protocol on managing pain intensity and functional disability in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Out of 70-millions older adults in the America, the majority of females have been suffering from osteoarthritis (OA) that progressively lead to chronic pain, joint stiffness, reduced mobility, muscle atrophy, poor balance, and ultimately, physical disability. Other physiological changes such as reduction in quadriceps' muscle strength and range of motion (ROM) in sagittal plane, and shortening of soft tissues around the joints collectively yield the distinctive clinical features such as articular pain; worsening on weight -bearing activities, resting/morning joint stiffness, progressive decline in physical activities and increasing to deformities/disabilities.Researchers observed the effectiveness of a structured exercise programs including an aerobic exercise program, a resistance exercise program, and a health education program in improving functional outcomes (self-reported disability) and decreasing the knee pain among older adults with knee OA at short-term and long term.the manual therapy along with supervised exercise protocol revealed a significant reduction in joint stiffness and knee pain and improvement in functional status of the patients with knee OA for short-term and long-term (1-year follow-up) than the placebo therapy (sub-therapeutic dose of ultrasound).

The study based on a randomized, pretest-posttest experimental group design, included a total of 32-participants with knee osteoarthritis randomly divided into groups A and B. Group A received a supervised exercise protocol, however group B received specified manual therapies in a combination of a supervised exercise protocol. Pain and functional disability measured with NPRS and WOMAC index respectively. Data collected on day-1st pre-intervention (baseline), day-14th posttest, and day-28th follow-up and analyzed using t-test and one-way ANOVA by keeping the level of significance at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* aged between 47 to 60 years;
* mild to moderate pain in one/both knees for 3-months;
* the pain intensity score between 2 to 6 on NPRS;
* morning stiffness <30-minutes;
* Self-reported crepitus on knee motion;
* grade 1 to 3 on Kellgren-Lawrence radiographic grading scale for Knee OA

Exclusion Criteria:

* diagnosed case of post-traumatic knee stiffness;
* history of bone infection and malignancy (osteomyelitis and tumour); neurological disorder (sciatica);
* history of joint replacement/meniscal surgery/mechanical knee pain/infection to the knee joint; suffering from severe cardiopulmonary disease (chronic obstructive pulmonary disease);
* Patient showed non-cooperation

Ages: 47 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 4-weeks
  Assessed by Numeric Pain Rating Scale (NPRS)
Functional disability | 4-weeks
  Assessed by WOMAC index

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT-Ortho, Principal Investigator — Rehabilitation Research Chair, CAMS, King Saud University, Riyadh, Saudi Arabia
Locations (1):
- Rehabilitation Research Chair, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No